CLINICAL TRIAL: NCT05917756
Title: The Impact of Mobilization With Movement on Pain, Function, and Quality of Life in Patients With Thoracic Outlet Syndrome: A Randomized Controlled Trial
Brief Title: Mobilization With Movement on Pain, Function, and Quality of Life in Patients With Thoracic Outlet Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ahram Canadian University (Other)
Responsible Party: Principal Investigator, Mohamed Magdy ElMeligie, Lecturer of Physical Therapy and Director of Electromyography Lab, Ahram Canadian University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 012/0333666
Record Dates: First submitted 2023-06-15; First posted 2023-06-26 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Thoracic Outlet Syndrome
MeSH Terms: conditions — Thoracic Outlet Syndrome | interventions — Movement

STUDY DESIGN:
Intervention Model Description: Two-arm randomized controlled trial with an equal allocation ratio (1:1) for the experimental and control groups
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (experimental group) (Experimental): MWM techniques combined with a tailored therapeutic exercise program
  Interventions: Other: Mobilization with Movement (MWM) and Tailored Therapeutic Exercise Program
- Group B (control group) (Active Comparator): Conventional physiotherapy combined with a tailored therapeutic exercise program
  Interventions: Other: Conventional Physiotherapy

INTERVENTIONS:
Other: Mobilization with Movement (MWM) and Tailored Therapeutic Exercise Program — The intervention consists of MWM techniques targeting the cervical and thoracic spine, and the first rib, applied by a certified physiotherapist for 8 weeks, 2 sessions per week, each session lasting 45 minutes. The intervention also includes a tailored therapeutic exercise program for the patients, comprising postural correction, stretching, and strengthening exercises. This intervention will be compared to conventional physiotherapy in the control group.
  Arms: Group A (experimental group)
Other: Conventional Physiotherapy — Conventional physiotherapy, including manual therapy (soft tissue mobilization, joint mobilization, and nerve gliding techniques) for 8 weeks, 2 sessions per week, each session lasting 45 minutes, combined with a tailored therapeutic exercise program (including postural correction, stretching, and strengthening exercises).
  Arms: Group B (control group)

SUMMARY:
This randomized controlled trial aims to evaluate the effects of Mobilization with Movement (MWM) on pain, function, and quality of life in patients with Thoracic Outlet Syndrome (TOS) compared to conventional physiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-65 years, diagnosed with TOS by a specialist, and experiencing symptoms for at least 3 months

Exclusion Criteria:

* Previous surgery for TOS
* contraindications to manual therapy
* other comorbidities significantly affecting upper limb function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Changes in Pain Intensity | Changes in Pain intensity at Baseline, 4 weeks, 8 weeks, and 12 weeks (follow-up)
  Pain intensity will be assessed using the Numeric Pain Rating Scale (NPRS).

SECONDARY OUTCOMES:
Changes in Functional Status | Changes in Functional Status Baseline, 4 weeks, 8 weeks, and 12 weeks (follow-up)
  Functional status will be evaluated using the Disabilities of the Arm, Shoulder, and Hand (DASH) questionnaire.
Changes in Cervical Range of Motion | Baseline, 4 weeks, 8 weeks, and 12 weeks (follow-up)
  Cervical range of motion will be assessed using a goniometer.
Changes in Quality of Life | Changes in quality of life at Baseline, 4 weeks, 8 weeks, and 12 weeks (follow-up)aseline, 4 weeks, 8 weeks, and 12 weeks (follow-up)
  Quality of life will be assessed using the Short Form-36 (SF-36) questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Amal Fawzy, Ph.d, Study Director — Faculty of Physical Therapy, Ahram Canadian University
Locations (1):
- Outpatient clinic of faculty of physical therapy, Ahram Canadian University, Al Ḩayy Ath Thāmin, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No